CLINICAL TRIAL: NCT00068874
Title: Predictors of Adaptation and a Cognitive Behavioral Intervention for African American Adolescents With Lupus
Brief Title: Improving Quality of Life for African American Female Adolescents With Lupus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Ronald T. Brown, Ph.D., ABPP, Temple University, Department of Public Health
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P60AR049459 (NIH); P60AR049459 (NIH); NIAMS-094
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Lupus
Keywords: African American; Adolescent; Coping; Adjustment; Quality of Life
MeSH Terms: interventions — Coping Skills; Training Support

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Educational comparison group
  Interventions: Behavioral: Educational training
- 2 (Experimental): Group receiving coping intervention designed to enhance coping and psychological adjustment
  Interventions: Behavioral: Coping skills and cognitive restructuring techniques
- 3 (No Intervention): Comparison control group with no active intervention

INTERVENTIONS:
Behavioral: Coping skills and cognitive restructuring techniques — This is a cognitive psychoeducational program designed to enhance coping and adaptation to SLE. Participants will attend five study visits over 5 months. The first three visits are biweekly, 45-minute sessions during which the adolescent will be taught coping skills and cognitive restructuring techniques. The coping skills training will include training in relaxation, distraction, and problem-solving skills. The cognitive restructuring techniques will assist adolescents in using more accurate and adaptive cognitive responses.
  Other Names: HELP - Health Education for Lupus Patients
  Arms: 2
Behavioral: Educational training — Participants will attend five study visits that will include disease-appropriate education materials.
  Arms: 1

SUMMARY:
This study will evaluate a program designed to help African American adolescents with lupus (systemic lupus erythematosus or SLE) cope with the disease.

DETAILED DESCRIPTION:
SLE is the most common autoimmune connective tissue disease of childhood, affecting 5,000 to 10,000 children; the prevalence is higher among African American children and approximately 80% of sufferers are female. SLE is multisystemic in onset and has no known cure. Children with chronic illness have at least a two-fold increased risk for adjustment problems relative to their healthy peers. This risk is heightened among adolescents, who are at greater risk for psychopathology than are younger children. The diagnosis of a chronic medical condition during adolescence presents unique stressors, particularly for adolescents with lupus, who must endure bodily changes, including dermatological problems, hair loss, and changes in appearance due to medical therapies. Psychosocial processes, including methods of coping, expectations, and family functioning, are believed to mediate the influence of disease severity. This study will evaluate the effectiveness of a cognitive-based intervention to improve the quality of life of adolescents with SLE.

Participants in this study will be randomly assigned to either the cognitive-based intervention, a lupus education program, or a control group. Participants in the intervention group will have five study visits over 5 months. The first three visits are biweekly, 45-minute sessions during which the adolescent will be taught coping skills and cognitive restructuring techniques. The coping skills training will include training in relaxation, distraction, and problem-solving skills. The cognitive restructuring techniques will assist adolescents in using more accurate and adaptive cognitive responses. Caregivers will join the adolescent at the end of each training session to gain familiarity with the content reviewed in each session. The remaining two study visits are booster sessions during which the intervention material will be reviewed.

Participants in the education program will also have five study visits. Study visits will include disease-appropriate education materials. Caregivers will not be included in the education program. Participants will be assessed at study entry and Months 6, 9, and 12. Assessments will include questionnaires designed to measure disease severity, pain intensity, methods of coping, expectations of efficacy, social support, and adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic lupus erythematosus (SLE)

Exclusion Criteria:

* Severe depression with suicidal thoughts
* Delirium, dementia, or cognitive impairment (e.g., Mini Mental Status Examination 24 or less)
* Severe intellectual impairment
* Terminal illness with a life expectancy of less than 1 year

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
BASC scores (measures of general adjustment) | 4 years
BASS Scores | 4 years
SPPA scores (perception of physical appearance and social | 4 years
competence) | 4 years
Peds-QL 4.0 and 3.0 (quality of life assessments) | 4 years
Psychological Adjustment | 4 years
BASC Scores | 4 years

SECONDARY OUTCOMES:
SLEDAI (measure of disease status) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T. Brown, PhD, Principal Investigator — Department of Public Health - Temple University
Locations (1):
- Ronald T. Brown, PhD, Philadelphia, Pennsylvania, United States